CLINICAL TRIAL: NCT06585150
Title: A Phase 2 Randomized, Placebo-controlled Study of the Safety and Efficacy of Obeldesivir to Treat Nonhospitalized Adults With Acute Respiratory Syncytial Virus (RSV) Infection
Brief Title: Study of Obeldesivir to Treat Nonhospitalized Adults With Acute Respiratory Syncytial Virus (RSV) Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated by Sponsor; the decision was not due to any safety findings.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-685-6819
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: RSV Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Obeldesivir (ODV) (Experimental): Participants will receive obeldesivir for 5 days
  Interventions: Drug: Obeldesivir
- Placebo comparator: Obeldesivir Placebo (Experimental): Participants will receive obeldesivir placebo for 5 days
  Interventions: Drug: Obeldesivir Placebo

INTERVENTIONS:
Drug: Obeldesivir — Tablet administered orally
  Other Names: GS-5245
  Arms: Obeldesivir (ODV)
Drug: Obeldesivir Placebo — Tablet administered orally
  Arms: Placebo comparator: Obeldesivir Placebo

SUMMARY:
The goal of this clinical study is to learn more about the study drug, obeldesivir (ODV; GS-5245), and how safe and effective it is in treating nonhospitalized adults with acute respiratory syncytial virus (RSV) infection. The researchers want to see if obeldesivir can help participants' symptoms get better faster.

The primary objectives of this study are to evaluate the efficacy of ODV in reducing the duration of symptoms and to evaluate the safety and tolerability of ODV in nonhospitalized adult participants with acute RSV infection.

ELIGIBILITY:
Key Inclusion Criteria:

* Exhibits at least 1 of the following risk factors for severe RSV disease:

  1. Age ≥ 60 years
  2. Moderate or severe chronic obstructive pulmonary disease (COPD) with a history of exacerbation during the preceding 12 months.
  3. Asthma with a history of ≥ 1 exacerbation during the proceeding 12 months
  4. One or more of the following chronic lung diseases:

     * i) Bronchiectasis
     * ii) Interstitial lung disease (eg, idiopathic pulmonary fibrosis)
     * iii) Pulmonary hypertension
  5. Chronic cardiovascular disease exclusive of hypertension
* RSV infection confirmed ≤ 3 days before randomization
* New onset or increased from baseline of ≥ 2 of the following signs and or/symptoms, and at least 1 sign/symptom of moderate severity a screening, and onset ≤ 3 days before randomization.
* RSV vaccine status:

  * Individuals whose only risk factor is age ≥ 60 years must not have received any doses of a vaccine for RSV.

Key Exclusion Criteria:

* Currently requiring or expected to require hospitalization within 48 hours after randomization.
* Documented previous infection and/or hospitalization for RSV during the current respiratory virus season.
* Documented to be positive for influenza A or B virus, and/or severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) ≤ 7 days prior to randomization.
* Concurrent infections requiring treatment with any antimicrobial therapy ≤ 7 days prior to randomization.
* Individuals with a history of cystic fibrosis.
* Undergoing dialysis, known history of moderate or severe renal impairment within the preceding 6 months prior to randomization.
* Pregnant at screening.
* Received any approved or authorized, direct-acting antiviral drug or monoclonal antibody against RSV < 28 days or < 5 half-lives, whichever is longer, before randomization.
* Received an investigational product < 28 days or < 5 half-lives, whichever is longer, before randomization.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Time to Alleviation of Targeted Respiratory Syncytial Virus (RSV) Symptoms as Measured by Respiratory Infection Intensity and Impact Questionnaire (RiiQ) through Day 15 | Day 1 up to Day 15
  The RiiQ symptom scale is a 13-item questionnaire rated on a 4-point scale. Each symptom is rated on a scale of 0 to 3 where 0=None, 1=Mild, 2=Moderate, and 3=Severe. Higher scores indicated greater severity.
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) Through Day 29 | Up to 29 days
Percentage of Participants Experiencing Laboratory Abnormalities Through Day 29 | Up to 29 days
Percentage of Participants Experiencing Serious Adverse Events (SAEs) and Adverse Events (AEs) Leading to Study Drug Discontinuation | First dose date up to Day 60

SECONDARY OUTCOMES:
Time to Sustained Alleviation of Targeted RSV Symptoms as Measured by RiiQ Through Day 15 | Day 1 up to Day 15
  The RiiQ symptom scale is a 13-item questionnaire rated on a 4-point scale. Each symptom is rated on a scale of 0 to 3 where 0=None, 1=Mild, 2=Moderate, and 3=Severe. Higher scores indicated greater severity.
Time to RSV-Related Lower Respiratory Tract Infection (LRTI) Through Day 29 | Day 1 up to Day 29
  RSV-related LRTI will be defined by symptoms (eg, cough, shortness of breath, wheezing, expectoration [coughing up mucus]) as assessed by the RiiQ symptom scale.
Time to RSV-Related Hospitalization or all-Cause Death Through Day 29 | Day 1 up to Day 29
  RSV-related hospitalization is defined as ≥ 24 hours of acute care for a reason related to RSV, in a hospital or similar acute care facility, including emergency rooms or temporary facilities instituted to address medical needs of those with RSV.
Time to RSV-Related Medically Attended Visit (MAVs) or all-Cause Death Through Day 29 | Day 1 up to Day 29
Change from baseline in RSV Viral Load Through Day 3 | Baseline, Day 3
Change from Baseline in RSV Viral Load Through Day 5 | Baseline, Day 5
Change from Baseline in RSV Viral Load Through Day 7 | Baseline, Day 7
Change from Baseline in RSV Viral Load Through Day 10 | Baseline, Day 10
Change from Baseline in RSV Viral Load Through Day 15 | Baseline, Day 15
Pharmacokinetic (PK) Parameter: AUCtau of GS-441524 | Day 1 to Day 5
  AUCtau is defined as the area under the concentration versus time curve over the dosing interval.
PK Parameter: Ctrough of GS-441524 | Day 1 to Day 5
  Ctrough is defined as the concentration at the end of the dosing interval
PK Parameter: Cmax of GS-441524 | Day 1 to Day 5
  Cmax is defined as the maximum observed concentration of drug in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (120):
- United States (120):
  - Central Alabama Research, Birmingham, Alabama
  - Cullman Clinical Trials, Cullman, Alabama
  - Lakeview Clinical Research, LLC, Guntersville, Alabama
  - Headlands Research-Scottsdale, Scottsdale, Arizona
  - Epic Medical Research-Surprise, Surprise, Arizona
  - Clearview Medical Research, LLC, Canyon Country, California
  - Kaiser Permanente Fontana Medica Center, Fontana, California
  - University of California, San Francisco-Fresno, Fresno, California
  - Downtown L.A. Research Center, Inc., Los Angeles, California
  - L.A. Universal Research Center, INC., Los Angeles, California
  - Stanford, Palo Alto, California
  - National Institute of Clinical Research, Inc, Pomona, California
  - Paradigm Clinical Research, Redding, California
  - M3 Wake Research San Diego, San Diego, California
  - FOMAT Medical Research - Central Coast Family Care, Santa Maria, California
  - Med Partners, Inc., Toluca Lake, California
  - Allianz Research Institute- Colorado, Aurora, Colorado
  - Paradigm Clinical Research Centers, LLC., Wheat Ridge, Wheat Ridge, Colorado
  - Yale University, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Encore Medical Research of Boynton Beach, LLC, Boynton Beach, Florida
  - C & A Clinical trials Corp, Cape Coral, Florida
  - Prestige Clinical Research Center Inc, Coral Gables, Florida
  - Beautiful Minds Clinical Research Center, Cutler Bay, Florida
  - UHC Research, LLC, Doral, Florida
  - Dolphin Medical Research, Doral, Florida
  - Proactive Clinical Research, LLC, Fort Lauderdale, Florida
  - Aga Clinical Trials, Hialeah, Florida
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - Research In Miami, Inc., Hialeah, Florida
  - Doral Medical Research, LLC, Hialeah, Florida
  - Sync, LLC, Hialeah, Florida
  - Evolution Clinical Trials, Hialeah Gardens, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Health Awareness, LLC, Jupiter, Florida
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - Accel Research Sites - St. Pete-Largo Clinical Research Unit, Largo, Florida
  - Clinical Site Partners LLC dba Flourish Research, Leesburg, Florida
  - Angels Clinical Research Institute, Miami, Florida
  - LCC Medical Research Institute, Miami, Florida
  - CCM Clinical Research Group, LLC., Miami, Florida
  - Retreat Medical Research, Miami, Florida
  - Clinical Trial Services, Corp, Miami, Florida
  - Continental Clinical Research, LLC, Miami, Florida
  - Dynamic Medical Research, LLC - Miami, Miami, Florida
  - Nuren Medical & Research Center, Miami, Florida
  - Advanced Care and Clinical Trials, LLC, Miami, Florida
  - Cordova Research Institute, Miami, Florida
  - Miami Clinical Research, Miami, Florida
  - Research Institute of South Florida, Inc., Miami, Florida
  - P&S Research, LLC., Miami, Florida
  - Pro Live Medical Research, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Links Clinical Trials LLC, Miami, Florida
  - Reed Medical Research, Miami, Florida
  - Nuovida Research Center, Corp, Miami, Florida
  - Pro-Care Research Center, Miami Gardens, Florida
  - Essential Clinical Research, Inc, Miami Lakes, Florida
  - Southern Clinical Research, LLC, Miami Lakes, Florida
  - Oceanic Research Group, North Miami Beach, Florida
  - Palm Springs Community Health Center, Palm Springs, Florida
  - USPA Advance Concept Medical Research Group. LLC, South Miami, Florida
  - Angels Clinical Research Institute, Tampa, Florida
  - Precision Research Center Inc, Tampa, Florida
  - Santos Research Center, Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Encore Medical Research of Weston, Weston, Florida
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - Paradigm Clinical Research, Boise, Idaho
  - Clinical Research Prime, Idaho Falls, Idaho
  - Metro Infectious Disease Consultants, Burr Ridge, Illinois
  - Endeavor Health - Clinical Trials Center, Skokie, Illinois
  - University of Iowa, Iowa City, Iowa
  - Tranquil Clinical Research, Webster, Iowa
  - CCT Research- Versailles Family Medicine, Versailles, Kentucky
  - Centennial Medical Group, Columbia, Maryland
  - Great Lakes Research Institute, Southfield, Michigan
  - Javara Inc., Mankato, Minnesota
  - University of Minnesota, Saint Paul, Minnesota
  - Hannibal Regional Healthcare System, Inc, Hannibal, Missouri
  - Clay-Platte Family Medicine/Avacare, Kansas City, Missouri
  - Velocity Clinical Research, Lincoln, Nebraska
  - Be Well Clinical Studies, Lincoln, Nebraska
  - Velocity Clinical Research, Norfolk, Nebraska
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Prime Global Research, Inc., New York, New York
  - NYC Health and Hospitals-Lincoln, The Bronx, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - Eximia Research-NC, LLC, Raleigh, North Carolina
  - Wake Research, Raleigh, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - The Lidner Research Center at The Christ Hospital, Cincinnati, Ohio
  - Epic Medical Research- Oklahoma, Chickasha, Oklahoma
  - Velocity Clinical Research - Anderson, Anderson, South Carolina
  - Central Texas Clinical Research, Austin, Texas
  - Inquest Clinical Research, Baytown, Texas
  - PanAmerican Clinical Research, LLC, Brownsville, Texas
  - Epic Medical Research-Carrollton, Carrollton, Texas
  - WR- Global Medical Research, LLC, Dallas, Texas
  - Vilo Research Group, Inc, Houston, Texas
  - C & R Research Services USA, Inc., Houston, Texas
  - Diversified Medical Practices, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Santa Clara Family Clinic, Houston, Texas
  - Next Level Urgent Care, Houston, Texas
  - The Crofoot Research Center, INC., Houston, Texas
  - Helios Clinical Keller, Keller, Texas
  - Andres Garcia-Zuniga, MD, PA, Laredo, Texas
  - Metroplex Pulmonary and Sleep Center, McKinney, Texas
  - SMS Clinical Research, Mesquite, Texas
  - Epic Medical Research LLC - DeSoto, Red Oak, Texas
  - Medrasa Clinical Research, Sherman, Texas
  - Velocity Clinical Research-Salt Lake City, West Jordan, Utah
  - Velocity Clinical Research- Suffolk, Portsmouth, Virginia
  - Providence Regional Medical Center Everett, Everett, Washington
  - Swedish Organ transplant and Liver Center, Seattle, Washington
  - Frontier Clinical Research. LLC Kingwood, Kingwood, West Virginia
  - Frontier Clinical Research, LLC, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06585150